CLINICAL TRIAL: NCT05045521
Title: Comparison of Plyometric and Resistance Warmup on Running Performance in Recreational Athletes
Brief Title: Comparison of Plyometric and Resistance Warmup on Running Performance in Athlets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00850 Tehmina Gul
Record Dates: First submitted 2021-08-23; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Sports Physical Therapy
Keywords: Flexibility; Plyometric warm up; resistance warm up; running performance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- plyometric warm up group (Experimental): set of active exercises used as warm up protocol.
  Interventions: Other: plyometric warm up group
- resistance warm up group (Experimental): warm up protocol on treadmill wearing weighted jacket
  Interventions: Other: resistance warm up
- control (Active Comparator): warm up protocol on treadmill without weights
  Interventions: Other: control warm up group

INTERVENTIONS:
Other: plyometric warm up group — participants will be asked to do 10 minutes self-paced jog on motorized treadmill.
  During the plyometric intervention, subjects will perform the 2 * 8 squat jumps, 2 * 8 scissor jumps, and 2 * 8 double leg bounds (2 sets of 8 repetitions) as a part of warm-up, and will have 60 s to recover between each set. Prior to the intervention, participants will be shown the technique to be used during jumping through use of three videos.
  Arms: plyometric warm up group
Other: resistance warm up — participants will be asked to do 10 minutes self-paced jog on motorized treadmill.
  After the jog participants will perform the 6*10s strides with the 15% of the weight. Velocity of the strides will be controlled by the participants.
  Warmup will be followed by the 10minutes rest
  Arms: resistance warm up group
Other: control warm up group — participants will be asked to do 10 minutes self-paced jog on a motorized treadmill.
  After the jog participants will perform the 6*10s strides without the weight. Velocity of the strides will be controlled by the participants. Warmup will be followed by the 10minutes rest The total amount of time spended in each of the three warm-up protocols will be recorded. Participants will be instructed to wear the same pair of running shoes during the three tests.
  Arms: control

SUMMARY:
Background: Active Warm up is one of the best and commonly used techniques in athletes that can induce special type of cardiovascular and metabolic changes that can bring the prominent change in running performance. Warm up prepares the body to withstand the high intensity exercises and improves the athletic performance and reduce the risk of musculoskeletal injury.

Objective: The objectives of study are to compare two types of warm up resistance and plyometric warm up in recreational athletes to improve running performance.

DETAILED DESCRIPTION:
Warm up is initial practices before starting exercise with usual concept to enhance the overall performance generally known as warm up. Often prior to initiate specific sport it is recommended to do cardiovascular warm like stretching for at least 10 to 20 minutes. As believed by and proven to many sport coaches that warm up decline the risk of musculoskeletal injuries, improve player performance in particular sport by helps to upgrade body temperature, excel the muscle potential, decrease muscle stiffness as well as resistance, regulate muscle contractile units, increase heart rate and blood flow toward muscles, increase oxygen saturation, improve and regulate neuro-muscular electrical signals to achieve best outcome in competition.

Types of Warm Up:

Different types of warm up like active, passive and mixed regimes are generally recommended previous to any sport, different researches and studies have been conducted to seek the effects of various warm up protocols and their impact on athletes performance. Stretching, treadmill walking, plyometric exercises are frequently directed for warm up.

Plyometric warmup are heavy strength regimes may include works out like jumping, additionally called plyometric works out, ordinarily used to expand strength through the stretch-shortening cycle (SSC). This sort of preparing is a profoundly successful neuromuscular boost, with the benefit of requiring low physical space, time and it also require less training equipment to finish the training sittings. Present moment plyometric programs positively affect endurance running execution or running economy.

Resistance training improvement can improve running mechanics. Improved biomechanical efficiency and improved joint activation and coordination of leg muscles may enable a reduction in relative workload. Improved Running Mechanisms Combining neuromuscular efficiency and strength can reduce oxygen consumption and thus improve running economy and ultimately performance Indeed, the combination of HRT and plyometric training may facilitate further improvements in the running economy through the accumulation of adaptations previously observed when any type of training is run alone.

Previously investigated the effects of short term resistance training program and plyometric training on fitness performance in boys aged 12 to 15 years and concluded that plyometric training improved the running velocity. A study effect of plyometric training on running performance and vertical jumping in prepubertal boys it stated that plyometric training programme causes higher muscle tension compared to resistance training and energy is more stored and released during muscle shortening for this reason plyometric training is widely recommended for improving the running economy. A study was done on The Impact of Resistance Training on Distance Running Performance concluded that the running economy improved up to 8% with the help of resistance training programme but it improves the running performance in only trained runners. Even a small improvement in running economy could have a large impact on distance running performance, particularly in longer events, such as marathons or ultra-marathon. A study Effects of plyometric training on endurance and explosive strength performance in competitive middle- and long-distance runners.

ELIGIBILITY:
Inclusion Criteria:

* • Both male and female gender

  * Volunteers between age 19 to 25 years
  * Having total exercise load less than 5 hours per week
  * BMI having between 18.5kg/m2 to 25kg/m2
  * Must fulfill the 10 minutes' walk test on treadmill before starting the warmup (8).

Exclusion Criteria:

* • Any cardiovascular and neurological diseases,

  * Suffering from any musculoskeletal injuries; Any history of traumatic injuries

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Incremental Test. (Time of Exhaustion) | day 1
  Initial velocity will be 7 km h/1 and increased by 1 km h/1every 3 min up to 10 km h/1. The gradient of the motorized treadmill will be set at 1% to simulate the air resistance that athletes experience on an outdoor track. During the incremental test, at 10 km h/1, the gradient will be increased by 2.5% every 2 min until exhaustion. total distance and the time of exhaustion was noted.

SECONDARY OUTCOMES:
Modified Borg Scale (Rate of Perceived Exertion) | day 1
  The Borg rating of perceived exertion (RPE) scale developed by Swedish researcher Gunnar Borg is a tool for measuring an individual's effort and exertion, breathlessness and fatigue during physical work and so is highly relevant for occupational health and safety practice. In its simplest terms, it provides a measure of how hard it feels that the body is working based on the phys¬ical sensations that the subject experiences. the scale ranges from 0-10 with 0 at no exertion and 10 at maximum exertion.
Visual Analogue Fatigue Scale (VAFS) | day 1
  How effectively do you think the warm-up was in preparation for racing and requested to rate their readiness from 1 (not effective at all) to 10 (extremely effective). Please mark an "X" on the number line which describes your global fatigue with 0 being worst and 10 being normal.
Cardiopulmonary Yo- Yo Test. (Endurance Competition) | day 2
  The main objective of the Yo Y o test is to measure the ability to repeatedly perform intense exercise including the potential to rapidly recover from such exercise. During the Yo Yo test, participants perform repeated 2 × 20-m runs at progressively increasing speed, intermitted by 10-s periods of active recovery (2 × 5 m). The test is performed until total exhaustion of the participant is reached.
sargent jump test | day 1
  Ten mins rest after warm up sargent jump test for the determination of lower limb power the person jumps as high as he can for 3 times to reach at the highest distance on wall.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Aman Medical Institute, Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1) Ahsan M. A Comparative Study of Different Types of Warm-up Effect on Postural Stability and Isokinetic Strength. Indian Journal of Public Health Research & Development. 2019;10
- [Background] Ramirez-Campillo R, Alvarez C, Henriquez-Olguin C, Baez EB, Martinez C, Andrade DC, Izquierdo M. Effects of plyometric training on endurance and explosive strength performance in competitive middle- and long-distance runners. J Strength Cond Res. 2014 Jan;28(1):97-104. doi: 10.1519/JSC.0b013e3182a1f44c. PMID 23838975
- [Background] Ruben RM, Molinari MA, Bibbee CA, Childress MA, Harman MS, Reed KP, Haff GG. The acute effects of an ascending squat protocol on performance during horizontal plyometric jumps. J Strength Cond Res. 2010 Feb;24(2):358-69. doi: 10.1519/JSC.0b013e3181cc26e0. PMID 20072064
- [Background] Faigenbaum AD, McFarland JE, Keiper FB, Tevlin W, Ratamess NA, Kang J, Hoffman JR. Effects of a short-term plyometric and resistance training program on fitness performance in boys age 12 to 15 years. J Sports Sci Med. 2007 Dec 1;6(4):519-25. eCollection 2007. PMID 24149486
- [Background] Kotzamanidis C. Effect of plyometric training on running performance and vertical jumping in prepubertal boys. J Strength Cond Res. 2006 May;20(2):441-5. doi: 10.1519/R-16194.1. PMID 16686577
- [Background] Jung AP. The impact of resistance training on distance running performance. Sports Med. 2003;33(7):539-52. doi: 10.2165/00007256-200333070-00005. PMID 12762828
- [Background] Wei C, Yu L, Duncan B, Renfree A. A Plyometric Warm-Up Protocol Improves Running Economy in Recreational Endurance Athletes. Front Physiol. 2020 Mar 12;11:197. doi: 10.3389/fphys.2020.00197. eCollection 2020. PMID 32226393
- [Background] Lum D, Tan F, Pang J, Barbosa TM. Effects of intermittent sprint and plyometric training on endurance running performance. J Sport Health Sci. 2019 Sep;8(5):471-477. doi: 10.1016/j.jshs.2016.08.005. Epub 2016 Aug 17. PMID 31534822
- [Background] Grieco CR, Cortes N, Greska EK, Lucci S, Onate JA. Effects of a combined resistance-plyometric training program on muscular strength, running economy, and Vo2peak in division I female soccer players. J Strength Cond Res. 2012 Sep;26(9):2570-6. doi: 10.1519/JSC.0b013e31823db1cf. PMID 22105047
- [Background] Hurley BF. Effects of resistive training on lipoprotein-lipid profiles: a comparison to aerobic exercise training. Med Sci Sports Exerc. 1989 Dec;21(6):689-93. doi: 10.1249/00005768-198912000-00012. PMID 2696856
- [Background] Ryan AS, Ivey FM, Hurlbut DE, Martel GF, Lemmer JT, Sorkin JD, Metter EJ, Fleg JL, Hurley BF. Regional bone mineral density after resistive training in young and older men and women. Scand J Med Sci Sports. 2004 Feb;14(1):16-23. doi: 10.1111/j.1600-0838.2003.00328.x. PMID 14723783